CLINICAL TRIAL: NCT02836314
Title: Effect Of Platelet Rich Fibrin on the Healing of Periodontal Intrabony Defects Treated With Anorganic Bovine Bone Mineral: A Randomized Clinical and Radiological Study
Brief Title: Clinical and Radiological Effect Of Platelet Rich Fibrin on the Healing of Periodontal Intrabony Periodontal Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Yasemin Sezgin, Dr, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03/10-12
Record Dates: First submitted 2016-07-08; First posted 2016-07-19 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Periodontitis; Intrabony Periodontal Defect
Keywords: Anorganic bovine bone mineral;; Graft; Intrabony periodontal defect; platelet rich fibrin
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRF and ABBM (Experimental): Intervention: Anorganic Bovine Bone Mineral and Platelet Rich fibrin is applied to the periodontal intrabony defects
  Interventions: Other: Anorganic Bovine Bone Mineral and Platelet Rich Fibrin (PRF)
- Anorganic Bovine Bone Mineral (Active Comparator): Intervention: Anorganic Bovine Bone Mineral is applied to the periodontal intrabony defects
  Interventions: Other: Anorganic Bovine Bone Mineral (ABBM)

INTERVENTIONS:
Other: Anorganic Bovine Bone Mineral (ABBM) — In the control group, periodontal intrabony defects were treated with ABBM alone.
  Arms: Anorganic Bovine Bone Mineral
Other: Anorganic Bovine Bone Mineral and Platelet Rich Fibrin (PRF) — In the test group, periodontal intrabony defects were treated with ABBM and PRF combination.
  Arms: PRF and ABBM

SUMMARY:
The aim of this split mouth, single-center, controlled study is to compare the healing of intrabony defects treated with a combination of Anorganic Bovine Bone Mineral (ABBM)/Platelet Rich Fibrin (PRF) or Anorganic Bovine Bone Mineral alone. The hypothesis being tested in the study was that PRF would augment the regenerative effects of ABBM in human intrabony defects.

DETAILED DESCRIPTION:
Anorganic bovine bone mineral (ABBM) is extensively used in the treatment of intrabony defects. Platelet rich fibrin (PRF) is a new generation platelet concentrate with a simplified technique. Although there are some studies on the use of PRF in the treatment of intrabony defects, to date none of them evaluate its additive effects with ABBM. Therefore, a randomized, split mouth clinical trial was conducted to compare the healing of intrabony defects treated with a PRF/ABBM combination and to those obtained with ABBM alone. Using a split mouth design, 15 paired intrabony defects were randomly treated with either ABBM alone (control group) or with ABBM- PRF combination (test group). The following clinical parameters and radiographic measurements were recorded at baseline and six months postoperatively: plaque index (PI), gingival index (GI), probing depth (PD), gingival recession (GR), clinical attachment level (CAL), vertical bone loss, the depth of the defect and defect angle

ELIGIBILITY:
Inclusion Criteria:

* no systemic diseases;
* a good level of oral hygiene (OH) (plaque index<0.15);
* presence of two paired two-wall or three-wall intrabony defects with probing depth ≥6mm and an intrabony component ≥3mm as detected on radiographs; -no intrabony defects extending into the furcation area;
* tooth mobility ≤1;
* tooth and adjoining teeth testing vital and without symptoms or signs of endodontic involvement;
* tooth and adjoining teeth free of caries or inadequate restorations.

Exclusion Criteria:

* patients with compromised immune systems;
* pregnant and/or lactating women;
* patients taking any drug known to affect the periodontal status or affect the coagulation system
* smokers.

Ages: 38 Years to 61 Years | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level change: The distance from cemento-enamel junction to the depth of the sulcus recorded by a periodontal probe at baseline and 6 months postoperatively | baseline and 6 months

SECONDARY OUTCOMES:
Vertical bone loss change: Distance between cemento-enamel junction and base of the defect measured in standardized radiographs at baseline and 6 months postoperatively | Baseline and 6 months
Probing depth change: The distance from the gingival margin to the depth of the sulcus recorded by a periodontal probe at baseline and 6 months postoperatively | baseline and 6 months
Radiographic defect angle change: Using the function 'angle' the defect angle can be measured by assessing the two lines that represent the root surface of the involved tooth and the bone defect surface at baseline and 6 months postoperatively | baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Levent Taner, PhD, DDS, Study Director — Gazi University, Faculty of Dentistry, Department of Periodontology
Locations (1):
- Yasemin Sezgin, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes